CLINICAL TRIAL: NCT07376759
Title: Effects of Comfort Theory-Based Education on Dysmenorrhea, Menstrual Symptoms, Premenstrual Syndrome and General Well-Being Levels in University Students With Primary Dysmenorrhea
Brief Title: Primary Dysmenorrhea and Comfort Theory
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ordu University (Other)
Collaborators: Ordu University Scientific Research Projects Coordination Department (Unknown)
Responsible Party: Principal Investigator, Ebru Aydın, PhD Student, Ordu University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: ODU-SBE-EA-01
Record Dates: First submitted 2026-01-21; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Primary Dysmenorrhea
Keywords: primary dysmenorrhea; comfort theory; menstrual symptoms; premenstrual syndrome; general wellbeing; nursing
MeSH Terms: conditions — Premenstrual Syndrome

STUDY DESIGN:
Intervention Model Description: This study consisted of two groups: 40 intervention group members and 40 control group members.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Active Comparator): The intervention group will receive training based on Kolcaba's Comfort Theory.
  Interventions: Other: Comfort Theory-Based Education
- control group (No Intervention): The control group will not be subjected to any intervention.

INTERVENTIONS:
Other: Comfort Theory-Based Education — The training program will be conducted face-to-face and through oral instruction. Each training session will last 40 minutes. A total of three training sessions will be given, one per month, over a three-month period.
  Arms: intervention group

SUMMARY:
Dysmenorrhea is defined as lower abdominal pain experienced during menstruation. It is divided into two types: primary dysmenorrhea and secondary dysmenorrhea. In young women, the majority of dysmenorrhea cases are primary dysmenorrhea. Primary dysmenorrhea has a physical, psychological, and social impact on young women. Pharmacological and non-pharmacological methods are used to treat primary dysmenorrhea. Education is important in increasing the effectiveness of primary dysmenorrhea treatment. An effective education process takes place in accordance with nursing theories and models. There are a limited number of studies on the effect of comfort theory-based education in the management of primary dysmenorrhea. In this research, planned as a randomized controlled trial, the intervention group will receive comfort theory-based education, while the control group will receive no intervention. This study aims to contribute to the literature by investigating the effect of comfort theory-based education on dysmenorrhea, menstrual symptoms, premenstrual syndrome, and general well-being in university students with primary dysmenorrhea.

ELIGIBILITY:
Inclusion Criteria:

* Female students aged 18 and over
* Single
* Having a menstrual pain intensity of 3 or higher according to the Visual Analog Scale
* Having had a regular menstrual cycle for the last 6 months
* Volunteering to participate in the study

Exclusion Criteria:

* Women diagnosed with a psychiatric illness
* Women diagnosed with a gynecological illness
* Women diagnosed with a chronic illness
* Women using a pharmacological or non-pharmacological method for primary dysmenorrhea
* Women using hormonal birth control methods

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale | three months
  On a scale consisting of a ruler, one end is marked "0" (the point where there is no pain) and the other end is marked "10" (the point where the pain is most severe). Pain levels are classified as follows: less than 3 is mild, 3-6 is moderate, and more than 6 is severe.

SECONDARY OUTCOMES:
Menstruation Symptom Scale | three months
  This scale consists of 22 items. Participants are asked to rate their menstrual symptoms on a scale of 1 (never) to 5 (always). The lowest score on the scale is 22, and the highest score is 110. A higher score indicates an increase in the severity of menstrual symptoms.
Dysmenorrhea Impact Scale | three months
  This scale consists of 13 items. Participants are asked to rate each item on a scale of 1 to 5. The lowest score on the scale is 13, and the highest score is 65. As participants' scores on the scale increase, their level of being affected by dysmenorrhea also increases.
Premenstrual Syndrome Scale | three months
  This scale consists of 44 items. Participants are asked to rate each item on a scale of 1 to 5. The lowest score is 44, and the highest score is 220. Higher scores indicate a higher severity of premenstrual syndrome
General Well-being Scale | three months
  This scale consists of 14 items. Participants are asked to rate each item on a scale of 1 to 5. The lowest score on the scale is 14, and the highest score is 70. As participants' scores on the scale increased, their overall level of well-being also increased.

IPD SHARING:
Plan to Share IPD: No